CLINICAL TRIAL: NCT05129878
Title: Effect of COCs Ethinylestradiol/Norethisterone Acetate Along With Scaling on Periodontal Health and hsCRP in Polycystic Ovary Syndrome Women Having Gingivitis : A Randomized Controlled Trial
Brief Title: Effect of EE/NETA With Scaling on Periodontium and hsCRP in PCOS Women With Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RICHA PERIO
Record Dates: First submitted 2021-08-22; First posted 2021-11-22 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Gingivitis; PCOS
MeSH Terms: conditions — Gingivitis | interventions — Tooth Exfoliation; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1 (Experimental): patients with PCOS on combined oral contraceptives (COCs) having gingivitis will receive scaling and oral hygiene instructions (OHI)
  Interventions: Procedure: scaling and OHI
- Test group 2 (Experimental): patients with PCOS on combined oral contraceptives (COCs) having gingivitis will receive oral hygiene instructions only
  Interventions: Procedure: oral Hygiene instructions
- Control Group (Active Comparator): Systemically Healthy (age and BMI matched) females with gingivitis will receive with OHI and scaling.
  Interventions: Procedure: Scaling and oral hygiene instruction

INTERVENTIONS:
Procedure: scaling and OHI — patients with PCOS on combined oral contraceptives (COCs) having gingivitis will receive scaling and oral hygiene instructions
  Arms: Test group 1
Procedure: oral Hygiene instructions — patients with PCOS on combined oral contraceptives (COCs) having gingivitis will receive oral hygiene instructions only
  Other Names: Education and motivation
  Arms: Test group 2
Procedure: Scaling and oral hygiene instruction — Systemically Healthy (age and BMI matched) females with gingivitis will receive with OHI and Scaling
  Arms: Control Group

SUMMARY:
As gingivitis is known to add to the systemic inflammatory burden and may consequently contribute to progression of PCOS and vice-versa, So, controlling local and systemic inflammatory burden by scaling g and medical treatment may have an effect in the management of PCOS women having gingivitis.There is no data as yet, comparing the impact of COCs along with scaling and COCs along with just oral hygiene instructions on the periodontal health of PCOS patients. Therefore, there is need to study the effect of combined oral contraceptives (ethinylestradiol/norethisterone acetate) along with scaling on periodontal status and high sensitivity C-Reactive Protein in polycystic ovary syndrome women having gingivitis

DETAILED DESCRIPTION:
Various studies have been conducted to assess the impact of oral contraceptives on periodontal status and mostly present conflicting results. However, none of these studies have been carried out on females diagnosed with PCOS. Such an assessment is significant keeping in mind the increasing prevalence of PCOS as well as introduction of low-dose oral contraceptives for the long-term management of these patients. Additionally, gingivitis is known to increase the systemic inflammatory burden and may possibly contribute to progression of PCOS and vice-versa. So, controlling both local and systemic inflammatory burden by scaling along with medical treatment may have a vital role in the management of PCOS women having gingivitis. There is no data as yet, evaluating the impact of COCs on the periodontal health of PCOS patients. Therefore, the effect of hormone based medical treatment on the periodontal status of these patients, whether protective or destructive, remains unclear till date. The present study, thus, aims to evaluate the effect of combined oral contraceptives (ethinylestradiol / norethisterone acetate) with and without scaling on the periodontal status and the levels of serological marker of inflammation {high sensitivity-C Reactive Protein (hsCRP)} among polycystic ovarian syndrome (PCOS) women having ginigvitis.

MATERIAL AND METHODOLOGY STUDY DESIGN AND SETTING- The present randomised controlled clinical trial will be conducted in the Department of Periodontology, Post Graduate Institute of Dental Sciences, Rohtak in collaboration with Department of Obstetrics and Gynecology, Post Graduate Institute of Medical Sciences, Rohtak.

STUDY PERIOD- 12-14 months STUDY SUBJECTS- PCOS patients having gingivitis,15-40 years of age and systemically healthy patients with gingivitis All the participants will be age and BMI matched. The present Randomized Controlled Trial will include 60 individuals of PCOS who will be divided into 2 groups using randomisation software. Generating randomization table.and allocation will be concealed in opaque envelops by another person not involved in the trial.30 systemically healthy females,age and BMI matched, will also be included.

Test group 1 , n=30, patients with PCOS on combined oral contraceptives (COCs) having gingivitis will receive oral hygiene instructions (OHI) and Scaling.

Test group 2, n=30, patients with PCOS on combined oral contraceptives (COCs) having gingivitis will receive oral hygiene instructions only Control Group , n=30, Systemically Healthy (age and BMI matched) females with gingivitis will receive with OHI and scaling.

Periodontal and anthropometric parameters will be measured and sampling will be done at baseline, 3months and 6 months. serum hsCRP levels will be assessed at baseline and at 6 months.

TEST GROUP AND CONTROL GROUPS - Periodontal parameters: -

1. PLAQUE INDEX
2. GINGIVAL INDEX
3. BLEEDING ON PROBING
4. GINGIVAL BIOTYPE
5. GINGIVAL RECESSION
6. ANALYSES OF ANTHROPOMETRIC PARAMETERS- Waist circumference (WC) waist-to-hip ratio (WHR) BMI(Kg/m²)
7. hsCRP LEVELS
8. PCOSQ (Polycystic ovary syndrome questionnaire)
9. ORAL HEALTH RELATED QUALITY OF LIFE (OHRqol) questionnaire
10. Phenotype of PCOS

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data recorded will be processed by standard statistical analysis.The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. If it is in normal distribution inter group comparison will be done by using Independent T test and paired t test will be use for intragroup comparison and if non-normal distribution of data, inter group comparison will be done by Mann-Whitney U test and intragroup by signed rank test. The Chi square test will be applied to analyze categoric data. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion Criteria:

- For test groups

* females of reproductive age group (15-40 yrs)
* BMI (18.5 - 24.9)
* The diagnosis of PCOS according to Rotterdam criteria(37), when any two out of the following three abnormalities will be present:

clinical (hirsutism, acne or acanthosis nigricans) and/or biochemical (raised testosterone) hyperandrogenism chronic anovulation (oligomenorrhoea or amenorrhea) polycystic ovaries on ultrasound (one or both ovaries demonstrate 12 or more follicles measuring 2 to 9 mm in diameter or the ovarian volume exceeds 10 cubic cm on pelvic ultrasound)

* presence of ≥20 natural teeth
* gingivitis by using the criteria laid down by World Workshop 2017

For Test Group 2

* Participants will receive professional oral hygiene instructions during the trial and will be given cause related treatment after observation period of 6 months.
* Delaying treatment will not be considered unethical because of the low risk of disease progression over 6 months (41) and because these individuals will be monitored frequently and offered immediate (rescue) treatment if their disease progresses. Such cases will be excluded from the study. Periodontitis progression will be defined as an increase in CAL of 2 mm at any tooth site(42).
* Participants will be enrolled in the present study after obtaining written informed consent after explaining the details of the study design in their native language.
* Also, patients with periodontitis or molar incisor pattern of periodontitis (2017 criteria) will not be included in the study For control group Systemically healthy females (age and BMI matched with PCOS women) diagnosed on the basis of regular menstruation, no clinical or biochemical sign of hyperandrogenism and ultrasound exclusion of PCOS, having gingivitis.

Exclusion Criteria:

* • history of androgen-secreting tumors, congenital adrenal hyperplasia and thyroid dysfunction

  * nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, active cancer within the last past 5 yrs
  * smokers and alcoholics
  * history of systemic antibiotics or oral contraceptives usage within last 3 months
  * periapical pathology or oral inflammatory conditions other than periodontitis.
  * any periodontal treatment within 6 months prior to study
  * incisor molar pattern/grade C periodontitis (2017 classification)

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 6 months
  BOP will recorded as 1 (present) if it occurred within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as % sites with bleeding on probing.
Serum high sensitivity C reactive protein (hsCRP) levels | 6 months
  Venous blood from the antecubital vein will be collected after applying a tourniquet in plain tubes without additive. Serum hsCRP levels will be assessed using a kit with high sensitivity methodology in an auto-analyzer according to the manufacturer's instructions. The test principle will be particle-enhanced immune-turbidimetric assay,in which human CRP agglutinates with the latex particles coated with monoclonal anti-CRP antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: RICHA VERMA, Principal Investigator — Post Graduate Institute of Dental Sciences,ROHTAK,HARYANA
Locations (2):
- India (2):
  - Post Graduate Institute of Dental Sciences, Rohtak, Haryana
  - Shikha Tewari, Rohtak, Haryana